CLINICAL TRIAL: NCT04357626
Title: Determinants of Rehabilitation Outcomes in Survivors of Primary Subarachnoid
Brief Title: Determinants of Rehabilitation Outcomes in Survivors of Primary Subarachnoid Haemorrhage
Acronym: DETERMINESAH
Status: Completed | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DSRB 2019/00594
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Subarachnoid Hemorrhage, Spontaneous
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Completed discharged hospital rehabilitation electronic record: Completed discharged hospital rehabilitation electronic record of patients who underwent inpatient rehabilitation as part of routine clinical care.
  Interventions: Other: Inpatient Rehabilitation

INTERVENTIONS:
Other: Inpatient Rehabilitation — Observational electronic records review study during inpatient rehabilitation

SUMMARY:
A retrospective, observational single centre study of electronic medical records of discharged patients who were admitted to from 1 January 2015 to 31 December 2018.

Period of data collection was from 5 August 2019 to 15 September 2019.

DETAILED DESCRIPTION:
The objectives of this study were to describe a local cohort of acute SAH survivors during inpatient rehabilitation at a single tertiary rehabilitation centre in Singapore and identify early predictors impacting discharge rehabilitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Spontaneous, first-ever SAH diagnosed by admitting neurosurgeons and confirmed on neuroimaging (CT or magnetic resonance imaging) 2. Transferred from acute care facilities or admitted from clinics to TTSH RC 3. Ages between 21 - 85 years 4. Duration of SAH to rehabilitation admission ≤6 months

Exclusion Criteria:

* 1. No radiological evidence of SAH 2. Traumatic SAH 3. Previous diagnosis of SAH 4. Main reason for admission into TTSH RC was not for inpatient rehabilitation (e.g. wound care, medical or social admission)

Ages: 21 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted acutely for inpatient rehabilitation from neurosurgical wards
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM score) | Within 72 hours of discharge from rehabilitation
  The FIM, scored between 18 - 126, comprises of 18 items (motor and cognitive sub scores) which assesses a patient's degree of disability and indicates the degree of assistance required for activities of daily living. FIM scoring is widely used for functional scoring in patients with neurologic pathologies such as stroke or traumatic brain injury. Studies on its utility have shown high reliability, validity, and sensitivity for measuring functional ability and high consistency with other functional scales such as the Barthel Index

SECONDARY OUTCOMES:
FIM Change | Within 72 hours of admission and discharge from rehabilitation
  Difference between FIM discharge and admission

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Chua, MBBS FRCPE, Principal Investigator — Tan Tock Seng Hospital
Locations (2):
- Singapore (2):
  - Tan Tock Seng Hospital, Singapore
  - Tan Tock Seng Hospital Rehabilitation Centre, Singapore

IPD SHARING:
Plan to Share IPD: No